CLINICAL TRIAL: NCT07134322
Title: From Conflict to Family Trauma - A Longitudinal Research for the Development of Best Practices in the Italian Legal System
Brief Title: From Conflict to Family Trauma
Acronym: FamilyTrauma
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lia Parente, Forensic Psychologist, University of Bari Aldo Moro
Other Study IDs: UniBa - UniSapienza
Record Dates: First submitted 2025-08-07; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Family Conflict; Family Characteristics; Family Dysfunctional
Keywords: Family Trauma; Higth Conflict; Therapeutic Jurisprudence
MeSH Terms: interventions — Hepatitis A Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study involves conflictual families who resort to the Court to restore parent-child relationship
  Interventions: Behavioral: The aim of this research is to record how many families go to court for the breakdown of parent-child relationships and to understand how many of these families, one year after the judge's ruling, hav

INTERVENTIONS:
Behavioral: The aim of this research is to record how many families go to court for the breakdown of parent-child relationships and to understand how many of these families, one year after the judge's ruling, hav — This is the first qualitative and quantitative study on conflict-ridden families who go to court and involve social and psychological support services.
  Furthermore, the survey will provide precise data on the extent of the phenomenon being investigated.

SUMMARY:
This project will examine the experience of the researcher as expert in the family court dealing with questions regarding family units, in conflict and children, victims of the family conflict, victims of abuse and neglect, often repeated over time.After the first consultation, family conflict often recurs, without regard for the treatment received, returning to the civil courts and sometimes to the criminal courts. There are three possibilities at this point, following the first decision of the court (a) there is a separation that resolves conflicts and leads to an improvement in outcomes for the children concerned; (b) pre-existing conditions specific to the children concerned continue, and the decision of the court regading separation has no effect; (c) conflict between the parents continues, with repeated returns to the civil courts, failure of processes of mediation and negotiation, and continuing or exacerbated trauma to the child leading to worse outcomes; (d) where there is a worse outcome, this may be due to the lack of supports following the expert psychological assessment and recommendation to the court..The forensic evaluation of the family often refers the family to public health services for therapeutic interventions and social supports. The lack of these interventions and supports of public health services may exacerbate the family trauma. This may occur (a) because the family conflict continues in the absence of the interventions and supports; (b) because the family trauma is exacerbated by continuing court proceedings because the conflict between parents concerning the care and placement of the children leads to prolonged legal proceedings and may result in worse outcomes for the children, such as criminal behaviour as this struggle continues. The child is 'instrumentalised', used as a pawn or weapon in the struggle between the parents. The research project aims first of all to outline, on the basis of the data to be acquired, (a) whether there is evidence that the decision of the court guided by the expert opinion and recommendations has a beneficial effect on outcomes for the child; (b) specific lines of treatment intervention and better packages of care and support to enhance good outcomes and minimise or prevent these adverse outcomes, under the supervision of the judge.

DETAILED DESCRIPTION:
This research project aims, to analyze the current practices and processes and to hypothesize possible support systems or the possibility of using existing resources with an element of training for clinicians, staff and experts.

Detailed Description This research project aims, to analyze the current practices and processes and to hypothesize possible support systems or the possibility of using existing resources with an element of training for clinicians, staff and experts.Furthermore, this research project aims to understand if certain characteristics of the members of the family unit or of the family unit as a system statistically influence the outcome of the treatment; understand if there is a need to create different support strategies for extreme conflict; to mobilise the support of lawyers, in order to actively involve them in the research project and together with the lawyers and the social services, find resolution strategies for this problem.

The project includes two phases of implementation:The first will concern, in agreement with the Ministry of Justice, the local public health and social services, the University and the Puglia Region Authority, the detection, starting from time T0 of all the family units that access the judicial system for the resolution of family disputes for which the assistance of an expert consultant is necessary to support the Judge in managing the dispute; this will include all the judicial offices belonging to the District of the Court of Appeal of Bari; the support will be sought of the specialist lawyers in the field who will join the research project and direct access to the files of the various Courts.This first phase, lasting a total of eighteen months, includes an initial period dedicated preliminarily to training/information on the data collection methods of the judicial office staff, jurists and experts of the public services involved in the research.

ELIGIBILITY:
Inclusion Criteria:

* Families with minor children who file a lawsuit
* Parent-child relationships must have been severed with at least one parent.

Exclusion Criteria:

- Families with adult children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All families in conflict with minor children who appear in court between January 2021 and December 2023 due to a breakdown in parent-child relationships.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-08 (Estimated); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of families with resolved conflict at 12 months | 1 year
  Data collection to determine whether, one year after the judge's ruling that found the parent-child relationship to be broken, the family conflict has been resolved and whether family ties have been restored. Specifically, through the court files of the Bari Court of Appeal district, the lawyers handling the case, and the public services appointed by the court to initiate the process of restoring family ties, we will identify how many family law cases, one year after treatment, have successfully resolved the issue of restoring the previously broken parent-child relationship and how many, however, remain unresolved.
  In particular:
  Time Frame: 12 months after baseline (T0) Description: Families in which the interventions indicated by the judge (e.g., mediation, therapy, parenting support) resulted in the resolution of parental conflict, confirmed by the absence of further court proceedings.
  Unit of Measure: Number of families
Number of children no longer involved in family conflict at 12 months | 1 year
  To determine how many minors, one year later, are still involved in family conflict and how many of these minors have developed psychological problems related to the ongoing family conflict. This data will be collected by consulting the court files of the Bari Court of Appeal District, the lawyers participating in the research, and the public services that, at the judge's direction, have taken charge of the complex family situation.
  In particular:
  Time Frame: 12 months after baseline (T0) Description: Children who are no longer directly involved in parental conflict, demonstrated by restored relationships with both parents or stabilization of custody and living arrangements.
  Unit of Measure: Number of children

SECONDARY OUTCOMES:
Number of children with restored parent-child relationship at 12 months | 12 months
  Time Frame: 12 months after baseline (T0) Description: Children who re-established a functional relationship with the previously absent or rejected parent, which was the initial reason for the judicial proceeding.
  Unit of Measure: Number of children
Percentage of families complying with therapeutic or mediation recommendations at 12 months | 12 months after baseline (T0)
  Families who completed at least one of the interventions recommended by the judge (e.g., therapy, mediation, parenting programs).

IPD SHARING:
Plan to Share IPD: No